CLINICAL TRIAL: NCT06987266
Title: Establishment of Diagnosis and Classification System for Lung Interstitial and Airway Diseases (LIAD)
Acronym: EDCS-LIAD
Status: Not yet recruiting | Type: Observational
Sponsor: Xiangya Hospital of Central South University (Other)
Collaborators: Beijing Hospital (Other Government); Henan Provincial People's Hospital (Other); Zhejiang University (Other); Zhongshan Hospital (Xiamen), Fudan University (Other); The Affiliated Hospital of Qingdao University (Other); The Affiliated Hospital Of Guizhou Medical University (Other); China-Japan Friendship Hospital (Other); First Hospital of China Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: 20250507
Record Dates: First submitted 2025-05-07; First posted 2025-05-23 (Actual); Last update posted 2025-05-23 (Actual); Status verified 2025-05

CONDITIONS: Interstitial Lung Diseases (ILD); Airway Disease
MeSH Terms: conditions — Lung Diseases, Interstitial

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Biospecimen Retention: Samples Without DNA — sputum; alveolar lavage fluid; blood; urine; stool
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (7):
- COPD with ILA: Chronic obstructive pulmonary disease complicated with interstitial lung abnormalities: patients were treated routinely without additional intervention.
  Interventions: Other: no intervention
- PF with emphysema syndrome: Pulmonary fibrosis with emphysema syndrome: patients were treated routinely without additional intervention.
  Interventions: Other: no intervention
- NSIP: Nonspecific interstitial pneumonia: patients were treated routinely without additional intervention.
  Interventions: Other: no intervention
- IPF: Idiopathic pulmonary fibrosis: patients were treated routinely without additional intervention.
  Interventions: Other: no intervention
- COPD: Chronic obstructive pulmonary disease: patients were treated routinely without additional intervention.
  Interventions: Other: no intervention
- NSIP with airway disease: Nonspecific interstitial pneumonia with airway disease: patients were treated routinely without additional intervention.
  Interventions: Other: no intervention
- IPF with airway disease: Idiopathic pulmonary fibrosis with airway disease: patients were treated routinely without additional intervention.
  Interventions: Other: no intervention

INTERVENTIONS:
Other: no intervention — no ntervention

SUMMARY:
This study focuses on both hospitalized and outpatient populations. Through a multicenter, retrospective study, it aims to comprehensively characterize:The comorbidity of interstitial lung diseases (ILD) and airway diseases;The comorbidity of ILD with other intrapulmonary diseases;The comorbidity of airway diseases with other intrapulmonary diseases;The comorbidity of ILD and airway diseases with extrapulmonary diseases.Based on these findings, the study seeks to propose classification and diagnostic criteria for ILD and airway disease comorbidities.Additionally, a multicenter, prospective, disease-specific cohort study will be conducted to observe the prognosis of patients with ILD and/or airway diseases, identify prognostic factors, and grade the severity of comorbid conditions based on these factors.Finally, the study will analyze the current state of interventions and the medical costs associated with ILD and airway disease comorbidities through a cost-effectiveness analysis, aiming to propose new strategies for integrated disease management.

DETAILED DESCRIPTION:
This study is divided into two parts, the first part is a multi-center, retrospective study of 9 units in the past 12 months of medical records (10,000 cases) were analyzed; The second part is a multi-center, prospective, observational cohort study. A total of 900 patients with pulmonary interstitial and airway diseases were enrolled, including hospitalized patients, outpatients, and subjects to be confirmed for 2-year follow-up. The total study period was 4 years (2024 December to 2028 November) .

1. A retrospective study was conducted in 9 tertiary hospitals across the country to collect data on cases discharged from respiratory and critical care medicine departments in the previous 12 months (2024 February to February 2025)(about 10,000 cases) , from which cases with a diagnosis of interstitial lung disease, airway disease were screened according to the discharge diagnosis ICD-10 code (disease classification and Code National Clinical Edition 2.0)(Table 1) , the clinical data, chest CT, lung function and intervention measures of the cases were collected to describe the comorbidity and intervention situation of hospitalized pulmonary interstitial and airway diseases in our country, and to put forward the classification and diagnostic criteria of pulmonary interstitial and airway diseases.

   By collecting data on patients with interstitial lung disease and airway disease who had been hospitalized in the respiratory and critical care unit in the previous 12 months at 9 tertiary hospitals, to describe the distribution of diseases, treatment and medical burden of pulmonary interstitial and airway diseases, pulmonary interstitial diseases, airway diseases and other intrapulmonary diseases, pulmonary interstitial diseases, airway diseases and extrapulmonary diseases in hospitalized patients, etc. , the classification and diagnostic criteria of pulmonary interstitial and airway diseases were proposed.
2. A prospective cohort study of comorbidity pulmonary interstitial and airway diseases was conducted in 9 tertiary hospitals across the country. The cohort patients were from three sources, hospitalized in the department of respiratory and critical care medicine, and hospitalized in the department of respiratory and critical care medicine, or outpatient clinics and checkup centers. Part 1 and Part 2: Screening of COPD patients with and without interstitial lung disease, Idiopathic pulmonary fibrosis with and without airway disease, nonspecific interstitial pneumonia with and without airway disease, and pulmonary fibrosis with emphysema in the inpatient and outpatient departments of respiratory and critical care medicine. In the third part, patients with pulmonary interstitial and/or airway diseases requiring respiratory specialist diagnosis in the subject I physical examination population screening, and patients with pulmonary interstitial and/or airway diseases requiring treatment after specialist judgment, were included, the risk factors, clinical information and biological samples of the patients were collected and followed up for 2 years (once every 12 months) . The prognostic information of the patients was collected and the influencing factors related to the prognosis were identified. The severity of comorbidity pulmonary interstitial and airway diseases was graded by analyzing the prognostic factors. By analyzing the intervention status of pulmonary interstitial and airway comorbidity diseases and the cost-effectiveness of medical costs, a new strategy of co-management was proposed. At the same time, it provides data support for the research of the first, fourth, fifth and sixth topic, and provides biological sample support for the third topic.

Clinical data, healthcare resource use, and bio-specimens were collected at baseline and at 2-year follow-up (every 12 months) from 9 Grade III, Class A hospital of respiratory and critical care medicine inpatients, outpatients, and patients with specialty-diagnosed interstitial lung disease and airway disease in the subject 1 physical examination population, to conduct a multi-center, prospective cohort study of comorbidity pulmonary interstitial and airway diseases and identify the influencing factors related to the prognosis of patients with pulmonary interstitial and/or airway diseases. The severity of comorbidity pulmonary interstitial and airway diseases was graded by analyzing the prognostic factors. By analyzing the intervention status of pulmonary interstitial and airway comorbidity diseases and the cost-effectiveness of medical costs, a new strategy of co-management was proposed.

ELIGIBILITY:
Inclusion Criteria:

1. age between 40-80 years old;
2. inpatients with an admission diagnosis of COPD, Idiopathic pulmonary fibrosis, nonspecific interstitial pneumonia, patients with the following diagnoses were screened by chest CT (slice thickness ≤1.5 mm) during hospitalization and by in-hospital or prior pulmonary function;
3. the inpatients could complete pulmonary function and chest CT examination within 1 month after discharge;
4. among outpatients, patients with chronic obstructive pulmonary disease, idiopathic pulmonary fibrosis, nonspecific interstitial pneumonia, COPD with pulmonary interstitial abnormalities, idiopathic pulmonary fibrosis with airway lesions, nonspecific interstitial pneumonia with airway lesions, pulmonary fibrosis with emphysema syndrome were diagnosed through chest CT (layer thickness ≤1.5mm) and lung function;
5. provide informed consent.

Exclusion Criteria:

1. expected survival less than 12 months;
2. planned lung transplantation or pneumonectomy within 12 months;
3. pregnant or lactating women.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Among the inpatient or outpatient patients in 9 Grade A hospitals, 900 patients with COPD combined with/uncombined interstitial lung abnormalities, idiopathic pulmonary fibrosis combined with/uncombined airway disease, nonspecific interstitial pneumonia combined with/uncombined airway disease, pulmonary fibrosis combined with emphysema syndrome.
Sampling Method: Non-Probability Sample
Enrollment: 900 (Estimated)
Dates: Start 2025-05-20 (Estimated); Primary Completion 2028-11-30 (Estimated); Study Completion 2028-11-30 (Estimated)

PRIMARY OUTCOMES:
Number of acute exacerbation | 12 months，24 months
Annual rate/value of decline in lung function | 12 months，24 months
  The main indicators observed for the annual lung function decline rate include △FEV1/pred, △FVC/pred, △DLCO/pred, △FEF50%/pred, △FEF75%/pred, △MMEF/pred; the main indicators observed for the annual lung function decline value include △FEV1, △FVC, △DLCO
Survival status | 12 months，24 months
  questionnaire
Advances in chest imaging | 12 months，24 months
  Evaluation indicators of chest imaging advances include emphysema degree , airway wall thickness and Interstitial lung changes. Quantitative analysis of emphysema degree using Goddard score and FACT-Digital LungTM software. Quantitative analysis of airway wall thickness using FACT-Digital LungTM software (Pi10). Changes in lung interstitial mass were quantitatively analyzed using InferRead™ CT Lung mean log_jac.

SECONDARY OUTCOMES:
symptom assessment | 1 and 12 months, 24 months
  Symptom assessment was performed using mMRC scale
symptom assessment K-BILD scale | 1 and 12 months, 24 months
  Symptom assessment was performed using K-BILD scale
symptom assessment CAT scale | 1 and 12 months, 24 months
  Symptom assessment was performed using CAT scale

IPD SHARING:
Plan to Share IPD: No